CLINICAL TRIAL: NCT01140360
Title: Pilot Study of Gleevec/Imatinib Mesylate (STI-571, NSC 716051) in Neurofibromatosis (NF1) Patient With Plexiform Neurofibromas
Acronym: 0908-09
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Kent Robertson (Other)
Responsible Party: Sponsor-Investigator, Kent Robertson, Associate Professor of Pediatrics, Indiana University School of Medicine
Organization: Indiana University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NF/Gleevec DOD Trial; 0908-09 (Other: IUPUI IRB)
Record Dates: First submitted 2010-06-08; First posted 2010-06-09 (Estimated); Results first posted 2017-07-02 (Actual); Last update posted 2017-07-02 (Actual); Status verified 2017-06

CONDITIONS: Neurofibromatosis; Neurofibromas
Keywords: Neurofibromas
MeSH Terms: conditions — Neurofibromatoses; Neurofibroma | interventions — Imatinib Mesylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Gleevec (Experimental): Gleevec will be dosed orally with a starting dose of 100 mg twice daily for patients with a BSA > 1.8 m2 or 55 mg/m2 twice daily for patients with BSA < 1.8 m2. For patients with a BSA > 1.8 m2 the dose will increase by increments of 100 mg bid every two weeks as tolerated up to a maximum dose of 400 mg bid. For patients with a BSA < 1.8 m2 the dose will increase by increments of 55 mg/m2 bid every two weeks as tolerated up to a maximum dose of 220 mg/m2 bid.Treatment will continue for 6 months with an option to continue for 24 months if the patient is deriving a clinical benefit.
  Interventions: Drug: Gleevec

INTERVENTIONS:
Drug: Gleevec — Gleevec will be dosed orally with a starting dose of 100 mg twice daily for patients with a BSA > 1.8 m2 or 55 mg/m2 twice daily for patients with BSA < 1.8 m2. For patients with a BSA > 1.8 m2 the dose will increase by increments of 100 mg bid every two weeks as tolerated up to a maximum dose of 400 mg bid. For patients with a BSA < 1.8 m2 the dose will increase by increments of 55 mg/m2 bid every two weeks as tolerated up to a maximum dose of 220 mg/m2 bid.Treatment will continue for 6 months with an option to continue for 24 months if the patient is deriving a clinical benefit.
  Other Names: Imatinib Mesylate

SUMMARY:
This is a second Pilot Study to determine the efficacy of Gleevec® in neurofibromatosis (NF1) patients with plexiform neurofibromas using new response assessment modalities with the secondary goals of assessing Gleevec toxicity, and characterizing markers of response. The rationale for this study arises from the response of human and murine NF1 cells to Gleevec® in vitro, the response of a NF1 patient treated with Gleevec® for airway compression by a plexiform neurofibroma with a dramatic response not previously seen in NF1 therapy, and the experience in 37 NF1 patients treated with Gleevec® in the initial pilot study. Gleevec will be dosed orally with a starting dose of 100 mg twice daily for patients with a BSA > 1.8 m2 or 55 mg/m2 twice daily for patients with BSA < 1.8 m2. For patients with a BSA > 1.8 m2 the dose will increase by increments of 100 mg bid every two weeks as tolerated up to a maximum dose of 400 mg bid. For patients with a BSA < 1.8 m2 the dose will increase by increments of 55 mg/m2 bid every two weeks as tolerated up to a maximum dose of 220 mg/m2 bid. Treatment will continue for 6 months with an option to continue for 24 months if the patient is deriving a clinical benefit.

ELIGIBILITY:
Inclusion criteria

1. Patients > 3 years of age.
2. Diagnosis of neurofibromatosis type 1 (NF1).
3. Presence of clinically significant plexiform neurofibromas (biopsy proven if possible with tissue blocks available); defined as tumors that are potentially life threatening or are impinging on vital structures or significantly impair the quality of life from pain or other symptoms.
4. Patients must have measurable disease by magnetic resonance imaging (MRI).
5. Patients must have a Karnofsky of > 70% or Lansky of > 50% and a life expectancy of > 2 months.
6. Adequate end organ function, defined as the following:

   total bilirubin < 1.5 x ULN, SGOT and SGPT < 2.5 x UNL, creatinine < 1.5 x ULN, ANC > 1.5 x 109/L, platelets > 100 x 109/L.
7. Patients must be able to swallow whole pills.
8. Female patients of childbearing potential must have negative pregnancy test within 7 days before initiation of study drug dosing. Postmenopausal women must be amenorrheic for at least 12 months to be considered of non-childbearing potential. Male and female patients of reproductive potential must agree to employ an effective barrier method of birth control throughout the study and for up to 3 months following discontinuation of study drug.
9. Written, voluntary informed consent.

Exclusion criteria

1. Patient has received any other investigational agents within 28 days of first day of study drug dosing, unless the disease is rapidly progressing.
2. Patient is < 5 years free of another primary malignancy except: if the other primary malignancy is not currently clinically significant nor requiring active intervention, or if other primary malignancy is a basal cell skin cancer or a cervical carcinoma in situ. Existence of any other malignant disease is not allowed.
3. Patient with Grade III/IV cardiac problems as defined by the New York Heart Association Criteria. (i.e., congestive heart failure, myocardial infarction within 6 months of study)
4. Female patients who are pregnant or breast-feeding.
5. Patient has a severe and/or uncontrolled medical disease (i.e., uncontrolled diabetes, chronic renal disease, or active uncontrolled infection).
6. Patient has a known brain metastasis. Non-specific CNS changes on MRI/CT characteristic of NF1 are allowed, but not known CNS malignancies.
7. Patient has known chronic liver disease (i.e., chronic active hepatitis, and cirrhosis).
8. Patient has a known diagnosis of human immunodeficiency virus (HIV) infection.
9. Patient received chemotherapy within 4 weeks (6 weeks for nitrosourea or mitomycin-C) prior to study entry, unless the disease is rapidly progressing.
10. Patient previously received radiotherapy to greater than or equal to 25 % of the bone marrow
11. Patient had a major surgery within 2 weeks prior to study entry.
12. Patient with any significant history of non-compliance to medical regimens or with inability to grant reliable informed consent.
13. Patients who have or anticipate receiving permanent (or semi-permanent) metallic structures attached to their body. (e.g., braces on teeth, body piercings), which their physicians believe will interfere with the MRI.

Ages: 3 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2012-02; Primary Completion 2016-08 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kent Robertson, MD PhD, Principal Investigator — Indiana University
Locations (1):
- Riley Hospital for Children, Indianapolis, Indiana, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Gleevec
Started | 21
Completed | 15
Not Completed | 6

BASELINE CHARACTERISTICS:
Arm/Group | Gleevec
Number analyzed (Participants) | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 10
  Between 18 and 65 years | 11
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 20
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 19
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 21

OUTCOME MEASURES:

1. Primary Outcome: Disease Response
Description: To estimate the disease control rate (SD, PR, CR) with Gleevec/Imatinib Mesylate in patients with neurofibromas (NF1). The sum of the longest diameter (LD) for all target lesions will be calculated and reported as the disease measurement. Complete Response (CR) disappearance of target lesions. Partial Response (PR) at least a 30% decrease in the disease measurement, taking as reference the disease measurement done to confirm measurable disease at study entry. Progressive Disease (PD) at least a 20% increase in the disease measurement, taking as reference the smallest disease measurement recorded since the start of treatment. Stable Disease (SD) neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD taking as reference the smallest disease measurement since the treatment started.
Time Frame: 1 year
Population: 13 participants reached the 1 year evaluation time-point. 6 participants withdrew prior to the 1 year evaluation time-point.
Measure: Count of Participants; unit: Participants
Arm/Group | Gleevec
Number analyzed (Participants) | 13
Participants
  Stable Disease (SD) | 13
  Partial Response (PR) | 0
  Complete Response (CR) | 0
  Progressive Disease (PD) | 0

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Gleevec
Serious Adverse Events (participants affected / at risk) | 3/21
Other Adverse Events (participants affected / at risk) | 21/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gleevec (N=21)
Pseudoaneurysm of carotid artery (Vascular disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Hepatic Failure (Hepatobiliary disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gleevec (N=21)
alopecia (Skin and subcutaneous tissue disorders) | 2 (2)
Alanine aminotransferase increased (Investigations) | 3 (4)
Neutrophil count decreased (Investigations) | 7 (10)
anemia (Blood and lymphatic system disorders) | 9 (11)
anorexia (Metabolism and nutrition disorders) | 3 (3)
Aspartate aminotransferase increased (Investigations) | 3 (6)
Back Pain (General disorders) | 3 (4)
blood bilirubin increased (Investigations) | 3 (4)
hypocalcemia (Metabolism and nutrition disorders) | 2 (3)
Constipation (Gastrointestinal disorders) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 3 (5)
dizziness (Nervous system disorders) | 2 (2)
dysphagia (Gastrointestinal disorders) | 2 (3)
dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
edema limbs (General disorders) | 5 (6)
fatigue (General disorders) | 7 (9)
Headache (Nervous system disorders) | 6 (6)
puritits (Skin and subcutaneous tissue disorders) | 2 (2)
Lymphopenia (Blood and lymphatic system disorders) | 2 (4)
Nausea (Gastrointestinal disorders) | 10 (16)
Neck pain (Musculoskeletal and connective tissue disorders) | 3 (4)
hypokalemia (Metabolism and nutrition disorders) | 5 (9)
Urinary frequency (Renal and urinary disorders) | 3 (3)
vomitting (Gastrointestinal disorders) | 4 (4)
white blood cell decreased (Investigations) | 11 (16)
weight loss (Investigations) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes